CLINICAL TRIAL: NCT02360202
Title: Evaluation of Fluid Retention Due to Superpotent Topical Corticosteroid in Patients With Bullous Pemphigoid
Brief Title: Evaluation of Fluid Retention Due to Superpotent Topical Corticosteroid
Acronym: RECOPB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: 2014/110/HP; 2014-002804-26 (EudraCT Number)
Record Dates: First submitted 2015-01-07; First posted 2015-02-10 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Quartz Crystal Microbalance Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bullous pemphigoid patient treated with clobetasol propionate (Experimental): Impedance analysis in patient with bullous pemphigoid treated by Clobetasol Propionate cream treatment.
  Interventions: Procedure: Impedance analysis; Drug: Clobetasol Propionate cream treatment

INTERVENTIONS:
Procedure: Impedance analysis — Impedance analysis in patient with Bullous pemphigoid disease treated with clobetasol propionate.
  impedance analysis includes : fat measures, lean body mass, total body water, extracellular water phase angle
Drug: Clobetasol Propionate cream treatment — clobetasol propionate treatment initiated following French recommendations
  Other Names: DERMOVAL or CLARELUX cream

SUMMARY:
Clinical observation frequently shows a paradoxical effect of topical corticosteroids in charge of a sudden melting of edema in the first days of treatment, which could be due to mobilization of extracellular. No study has shown the value of this measure in patients treated with topical steroids. This uncertainty, coupled with the observation of the paradoxical effects of topical steroids on edema are some patients that despite the systemic absorption of clobetasol propionate, a salt-free diet is not currently recommended practice.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate whether there is fluid retention after introduction of clobetasol propionate treatment from 10 g/day dosage to 40 g / day in patients with bullous pemphigoid. Bio-impedance is a noninvasive device for measuring with an electric current of low intensity the different volumes of the human body. A preliminary experiment of impedance measurements in some patients with bullous pemphigoid (examination requested as part of a nutritional assessment) showed that these patients had mostly a total water loss without dehydration, corresponding to a significant undernutrition during 1 month of treatment, possibly related to muscle wasting and protein loss by skin erosions without obvious argument for fluid retention, justifying reproduce these measures on a larger number of patients and the other to accurately assess the evolution of nutritional parameters during the first month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age higher than 18
* Patient with bullous pemphigoid,
* Patient treated by local corticosteroid therapy (clobetasol propionate cream) but not yet processed or for less than 48 hours,
* Signed informed consent.
* Patient affiliated to Social Security Regimen
* Effective contraception in women of childbearing age (for postmenopausal women, confirmatory diagnosis of menopause will be collected)

Exclusion Criteria:

* Concomitant treatment with corticosteroids
* Recent introduction or recent (<6 weeks) treatment with diuretics, angiotensin-converting enzyme, receptor antagonist or anti-angiotensin renin (aliskiren)
* contraindication to the use of Clobetasol propionate (DERMOVAL and CLARELUX)
* Patient on salt diet (<or = to 5 g / d)
* Patients carry a defibrillator or a pace maker
* Amputated Patient
* Pregnant and lactating
* Patient with Urinary Incontinency
* Recent heart decompensation in the last 6 weeks
* known Nephrotic Syndrome
* known or Severe hepatic impairment
* Hypoalbuminaemia less than 20 g / l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in fluid retention at day 30 | Day 30
  Change from Baseline in extra-cellular water volume at day 30 measured by bioimpedance analysis

SECONDARY OUTCOMES:
Change from Baseline in fluid retention at day 7 | Day 7
  Change from Baseline in extra-cellular water volume at day 7 measured by bioimpedance analysis
Weight variation between day 1 and day 30 | Day 30
Urinary Sodium level variation between day 1 and day 30 | Day 30
Urinary creatinin level variation between day 1 and day 30 | Day 30
Brain Natriuretic Peptide level variation between day 1 and day 30 | Day 30
Change from Baseline in nutritional parameters at day 30 | Day 30
  bioimpedance analysis, C Reactive Protein level, albumin level, daily diet diary, Buzby index
Change from Baseline in bullous pemphigoid disease severity index at day 30 | Day 30
  BPDAI questionary assessment
Change from Baseline in bullous pemphigoid disease severity index at day 7 | Day 7
  BPDAI questionary assessment
Change from Baseline in corticoid administration dosage at days 30 | Day 30
  Evaluation of corticoid dosage between day 1 and day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Duvert Lehembre, Doctor, Principal Investigator — clinique dermatologique du chu de Rouen
Locations (1):
- Rouen University Hospital, Rouen, France